CLINICAL TRIAL: NCT05790057
Title: Subclinical Cardiovascular Changes in Patient With Non Alcoholic Fatty Liver Disease (Predictive Value of Speckle Tracking Echocardiography )
Brief Title: Subclinical Cardiovascular Changes in NAFLD Patient (Predictive Value of Speckle Tracking Echocardiography )
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Mohamed Magdy Eid, pricipal investigator , internal medicine resident, Assiut University
Other Study IDs: cardiac complication in NAFLD
Record Dates: First submitted 2023-02-21; First posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Liver Steatoses
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
the goal of this study (observational study ) is to learn about the subclinical cardiovascular changes in patients with nonalcoholic fatty liver . the main questions it aims to answer are

1. the role of speckle tracking echocardiogram in detection of subclinical cardiovascular complication in NAFLD patients
2. the role of fibroscan in diagnosis of nonalcoholic fatty liver the participant will be examined by fibroscan and speckle tracking echocardiogram

DETAILED DESCRIPTION:
The diagnosis of Non Alcoholic Fatty Liver Disease ( NAFLD) requires evidence of hepatic steatosis by either imaging or histology and the exclusion of secondary causes of hepatic fat accumulation such as use of medications e.g ( corticosteroids , amiodarone , methotrexate ) , hereditary disorders e.g ( Wilson's disease , alpha 1 antitrypsin deficiency ) or viral infections additionally daily alcoholic consumption mustn't exceed 30g for men and 20g for women 1 Nonalcoholic fatty liver disease is rising in prevalence along with levels of obesity and type 2 diabetes mellitus such that it is now the most common cause of chronic liver disease worldwide prevalence in general population is 25 to 30% but this rises to 70% in patients with obesity and type 2 diabetes mellitus.

Fibroscan is an evidence based ,transient elastography instrument for noninvasive evaluation of liver steatosis and fibrosis There are various studies substantiating the use of fibroscan in NAFLD. In a study by Wong et al 246 patients underwent liver stiffness measurement by fibroscan , In a study carried out by Yoneda et al , AUROC for F1 , F2 , F3 , F4 fibrosis were 0.881, 0.876 , 0.914 and 0.997 , respectively. Musso et al showed that for nonalcoholic steatohepatitis (NASH) with advanced fibrosis, , sensitivity and specificity of fibroscan were 0.85, 0.90 , 0.97 and 0.94 . Another study from India by sarin et al showed similar efficacy of fibroscan in NAFLD in patients from Northern India4 Convincing evidence now substantiates a strong association between the presence and severity of ( NAFLD) and the risk of cardiomyopathy (mainly left ventricular dysfunction and hypertrophy , possibly leading to heart failure and arrhythmias 5 Speckle-tracking Echocardiography a non-invasive ultrasound imaging technique allows an objective and quantitative evaluation of global and regional myocardial function independently from the angle of insonation and cardiac translational movements based on an analysis of the spatial dislocation of speckles on routine 2 dimensional sonograms Because of its potential benefits in the measurement of left ventricular function along with other systolic and diastolic echocardiographic parameters of left ventricular function measurement this novel technique is used in this study to assess the relationship between NAFLD and subclinical myocardial dysfunction

All participants will be subjected to full history and examination including :

* Demographic data with special habits
* Underlying comorbidity (Diabetes mellitus , Hypertension , Cardiovascular disease
* Symptoms of NAFLD eg: fatigue , loss of appetite , weight loss , pale stool
* Symptoms of cardiac dysfunction including eg :

  * heart failure ( shortness of breath , fatigue , swelling of the feet ankles ,legs , abdomen or neck veins )
  * arrhythmia ( fluttering feelings in the chest [palpitations} )
  * heart attack ( chest pain or discomfort upper back or neck pain , indigestion , heartburn , nausea or vomiting , extreme fatigue ,upper body discomfort , dizziness and shortness of breath )
* Therapeutic history eg : drugs causing NAFLD ( corticosteroids , antidepressants , antipsychotics ) antihypertensive drugs , drugs to control Diabetes mellitus , Antiarrhythmic & anti ischemic drugs
* EXAMINATION : *vital signs ( blood pressure , pulse , temperature , respiratory rate ) * dyslipidemic signs * cardiovascular examination chest examination * lower limb pulsation

  * Laboratory investigation including:

    1. liver function
    2. lipid profile
    3. HBA1C
    4. Renal function
    5. Erythrocyte sedimentation rate ( ESR) & C - Reactive protein test ( CRP)
  * Imaging including:

    1. Fibroscan :

       It is a special non-invasive ultrasound technology that measures liver stiffness (hardness) and fatty changes in the liver
    2. Ultrasonography
    3. Conventional Echocardiography :

       It is an imaging technique that enables accurate assessment of cardiac structures and cardiac function
    4. Speckle Tracking Echocardiography:
  * Study Scores including:

    1. ASCVD risk score (Atherosclerotic cardiovascular disease )
    2. CHA2DS2-VASc score

       * Sample size Sample size was calculated using Epi-Info7 based on prevalence of NAFLD and its subclinical cardiovascular abnormalities , the minimum patients required for this study is 60 patient
  * statistical analysis : statistical analysis will be performed using SPSS statistics ( statistical package for the social sciences) version 20 (USA) , patient characteristics and outcomes will be reported using standard descriptive statistics : frequency (percentage ) for categorical variables and mean (SD) continuous variables .

ELIGIBILITY:
Inclusion Criteria:

1. Patients above age of 18 years old
2. All patients showing degree of fibrosis and steatosis

   -

Exclusion Criteria:

* 1-Patients diagnosed with cardiac disease (previous or current )

  2-patients known to have chronic liver disease

  3-patients younger than 18 years old

  4-patients with hepatocellular cancer

  5-patients know to be alcoholic

  6-patients with previous history of hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: any patient above 18 years no specific gender is required , with no comorbidities ( not cardiac not hypertensive , no chronic liver disease , no hepatocellular carcinoma , not alcoholic
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
the sensitivity of fibroscan in diagnosis of NAFLD | baseline
  analysis of the results of fibroscan and test the sensitivity of fibroscan in measurement the degree of steatosis and diagnosis of NAFLD
role of speckle tracking echocardiogram in detection of subclinical cardiovascular complications of NAFLD | baseline
  speckle tracking echocardiogram will be used to to find any cardiac abnormality such as myocardial infarction , valvular diseases in NAFLD patients
comparison between conventional echocardiogram and speckle tracking echocardiogram in detection of subclinical cardiovascular complications of NAFLD patients | baseline
  comparison between the results and measurements of both conventional echocardiogram and speckle tracking echocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: lobna m abdelwaheed, professor, Study Director — supervisor of the research ( professor of internal medicine Assiut university; soheir m kasem, professor, Study Director — supervisor of the research ( professor of internal medicine Assiut university
Locations (1):
- Assiut university, Asyut, Assuit, Egypt

REFERENCES:
- [Background] Kasper P, Martin A, Lang S, Kutting F, Goeser T, Demir M, Steffen HM. NAFLD and cardiovascular diseases: a clinical review. Clin Res Cardiol. 2021 Jul;110(7):921-937. doi: 10.1007/s00392-020-01709-7. Epub 2020 Jul 21. PMID 32696080
- [Background] Newsome PN, Sasso M, Deeks JJ, Paredes A, Boursier J, Chan WK, Yilmaz Y, Czernichow S, Zheng MH, Wong VW, Allison M, Tsochatzis E, Anstee QM, Sheridan DA, Eddowes PJ, Guha IN, Cobbold JF, Paradis V, Bedossa P, Miette V, Fournier-Poizat C, Sandrin L, Harrison SA. FibroScan-AST (FAST) score for the non-invasive identification of patients with non-alcoholic steatohepatitis with significant activity and fibrosis: a prospective derivation and global validation study. Lancet Gastroenterol Hepatol. 2020 Apr;5(4):362-373. doi: 10.1016/S2468-1253(19)30383-8. Epub 2020 Feb 3. PMID 32027858
- [Background] Oeda S, Tanaka K, Oshima A, Matsumoto Y, Sueoka E, Takahashi H. Diagnostic Accuracy of FibroScan and Factors Affecting Measurements. Diagnostics (Basel). 2020 Nov 12;10(11):940. doi: 10.3390/diagnostics10110940. PMID 33198092
- [Background] Pathik P, Ravindra S, Ajay C, Prasad B, Jatin P, Prabha S. Fibroscan versus simple noninvasive screening tools in predicting fibrosis in high-risk nonalcoholic fatty liver disease patients from Western India. Ann Gastroenterol. 2015 Apr-Jun;28(2):281-286. PMID 25830783
- [Background] Anstee QM, Mantovani A, Tilg H, Targher G. Risk of cardiomyopathy and cardiac arrhythmias in patients with nonalcoholic fatty liver disease. Nat Rev Gastroenterol Hepatol. 2018 Jul;15(7):425-439. doi: 10.1038/s41575-018-0010-0. PMID 29713021
- [Background] Zamirian M MD, Samiee E MD, Moaref A MD, Abtahi F MD, Tahamtan M MD. Assessment of Subclinical Myocardial Changes in Non-Alcoholic Fatty Liver Disease: A Case-Control Study Using Speckle Tracking Echocardiography. Iran J Med Sci. 2018 Sep;43(5):466-472. PMID 30214098